CLINICAL TRIAL: NCT00527332
Title: General Anesthesia Versus Spinal Anesthesia Combined With Intrathecal Morphine in Abdominal Hysterectomy for Benign Gynecological Diseases. A Randomized Open Controlled Study.
Brief Title: Effects of General Anesthesia and Spinal-Morphine Anesthesia on Recovery and Comfort After Benign Abdominal Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Preben Kjolhede (Other)
Responsible Party: Sponsor-Investigator, Preben Kjolhede, Associate professor, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EudraCT nr 2006-002520-41
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Hysterectomy (MeSH nr: E04.950.300.399)
Keywords: Hospitalization; Postoperative care; Quality of Life; Health economy; Anesthesia. Spinal; Anesthesia, General
MeSH Terms: interventions — Bupivacaine; Morphine; Propofol; Fentanyl; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Spinal anesthesia combined with intrathecal morphine. Spinal anesthesia applied in intervertebral space L3/L4 or L2/L3 with hyperbaric bupivacaine 20 mg and morphine 0.2 mg intrathecally. Sedation with propofol.
  Interventions: Drug: Bupivacain; Drug: Morphine; Drug: Propofol
- B (Active Comparator): General anesthesia. General anesthesia induced with propofol, fentanyl and rocuronium, and maintained with propofol and oxygen in air. Rocuronium and fentanyl repeated when needed.
  Interventions: Drug: Propofol; Drug: Fentanyl; Drug: Rocuronbromid; Drug: Morphine

INTERVENTIONS:
Drug: Bupivacain — 5 mg/mL, 4 mL intrathecally as a single dos
  Other Names: Marcain spinal tung.; ATC-code: N01BB01
  Arms: A
Drug: Morphine — 0.4 mg/mL; 0.5 mL intrathecally as a single dosage
  Other Names: Morfin Special; ATC-code: N02AA01
  Arms: A
Drug: Propofol — 2-5 mg/kg body weight/hours IV (intravenously) for sedation during the surgery
  Other Names: ATC-code: N01AX10
  Arms: A
Drug: Propofol — Induction of anesthesia with 1-2 mg/kg body weight IV (intravenously). After intubation maintenance dosage of 6-10 mg/kg/hour IV during the surgery
  Other Names: ATC-code: N01AX10
  Arms: B
Drug: Fentanyl — 100-200 microgram IV (intravenously) at start of anesthesia. 50-100 microgram IV on demand during surgery.
  Other Names: ATC-code:N01AH01
  Arms: B
Drug: Rocuronbromid — 0.6 mg/kg body weight IV (intravenously) at induction of anesthesia. If additional muscle relaxation is needed during surgery 5-10 mg is injected IV. The drug is given only at induction of anesthesia and during surgery
  Other Names: Esmeron; ATC-code: M03AC09
  Arms: B
Drug: Morphine — 5 mg is given IV (intravenously) before end of surgery
  Other Names: ATC-code: N02AA01
  Arms: B

SUMMARY:
The purpose of this study is to determine whether spinal anesthesia combined with intrathecal morphine in abdominal hysterectomy on benign gynecological indications gives better outcome concerning duration of hospital stay and postoperative patient comfort than general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 60 years of age.
* Scheduled for abdominal hysterectomy - total or subtotal -on benign gynecological indication.
* At least one ovary planned to be preserved at the hysterectomy.
* Can understand and communicate in Swedish
* Accept participation after written and verbal information and after signed informed consent.
* Has supervision at home after discharge from hospital during the first couple of days and has access to a telephone.

Exclusion Criteria:

* Contra-indications against spinal or general anesthesia or the standard dosage of the study drugs
* ASA classification ≥ Class 3
* Postmenopausal women without HRT (hormone replacement therapy).
* Suspected gynecological malignancy
* Previously undergone bilateral oophorectomy
* Substantial physically disabled so that a normal recovery with early physical mobilization can not be anticipated.
* Mentally or severly psychic disabled

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Preben Kjölhede, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, University Hospital, Linköping; Lena Nilsson, MD, PhD, Study Director — Department of Anesthesiology, University Hospital, Linköping; Ninnie B. Wodlin, MD, Study Director — Department of Obstetrics and Gynecology, University Hospital, Linköping; Kenneth Krohn, MD, Principal Investigator — Department of Ostetrics and Gynecology, Vrinnevi Hospital, Norrköping; Lars Nordenberg, MD, Principal Investigator — Department of Anesthesiology, Vrinnevi Hospital, Norrköping; Mats D. Karlsson, MD, Principal Investigator — Department of Obstetrics and Gynecology, Ryhov Hospital, Jönköping; Veronica Annerhagen, MD, Principal Investigator — Department of Anesthesiology, Ryhov Hospital, Jönköping; Christina Gunnervik, MD, Principal Investigator — Department of Obstetrics and Gynecology, Värnamo Hospital; Magnus Trofast, MD, Principal Investigator — Department of Anesthesiology, Värnamo Hospital; Tomasz Stypa, MD, Principal Investigator — Department of Obstetrics and Gynecology, Eksjö Hospital; Albert Sundberg, MD, PhD, Principal Investigator — Department of Anesthesiology, Eksjö Hospital
Locations (5):
- Sweden (5):
  - Eksjö Hospital, Eksjö
  - Ryhov Hospital, Jönköping
  - University Hospital, Linköping
  - Vrinnevi Hospital, Norrköping
  - Värnamo Hospital, Värnamo

REFERENCES:
- [Background] Vårdtid, funktionskapacitet och sjukskrivningstider efter hysterektomi. Nationella data från 6503 patienter opererade år 2000 och 2001. Återrapport från Nationella registret för kvalitetsutveckling inom gynekologisk kirurgi (Gynop-registret), SFOG, 2003.
- [Background] Kehlet H, Wilmore DW. Multimodal strategies to improve surgical outcome. Am J Surg. 2002 Jun;183(6):630-41. doi: 10.1016/s0002-9610(02)00866-8. PMID 12095591
- [Background] Wilmore DW, Kehlet H. Management of patients in fast track surgery. BMJ. 2001 Feb 24;322(7284):473-6. doi: 10.1136/bmj.322.7284.473. No abstract available. PMID 11222424
- [Background] Moller C, Kehlet H, Friland SG, Schouenborg LO, Lund C, Ottesen B. Fast track hysterectomy. Eur J Obstet Gynecol Reprod Biol. 2001 Sep;98(1):18-22. doi: 10.1016/s0301-2115(01)00342-6. PMID 11516794
- [Background] Persson P, Wijma K, Hammar M, Kjolhede P. Psychological wellbeing after laparoscopic and abdominal hysterectomy--a randomised controlled multicentre study. BJOG. 2006 Sep;113(9):1023-30. doi: 10.1111/j.1471-0528.2006.01025.x. PMID 16956334
- [Background] Ellstrom MA, Astrom M, Moller A, Olsson JH, Hahlin M. A randomized trial comparing changes in psychological well-being and sexuality after laparoscopic and abdominal hysterectomy. Acta Obstet Gynecol Scand. 2003 Sep;82(9):871-5. doi: 10.1080/j.1600-0412.2003.00216.x. PMID 12911451
- [Derived] Kjolhede P, Langstrom P, Nilsson P, Wodlin NB, Nilsson L. The impact of quality of sleep on recovery from fast-track abdominal hysterectomy. J Clin Sleep Med. 2012 Aug 15;8(4):395-402. doi: 10.5664/jcsm.2032. PMID 22893770
- [Derived] Kjolhede P, Borendal Wodlin N, Nilsson L, Fredrikson M, Wijma K. Impact of stress coping capacity on recovery from abdominal hysterectomy in a fast-track programme: a prospective longitudinal study. BJOG. 2012 Jul;119(8):998-1006; discussion 1006-7. doi: 10.1111/j.1471-0528.2012.03342.x. Epub 2012 May 9. PMID 22568450

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Anesthesia: Spinal anesthesia combined with intrathecal morphine
- General Anesthesia: General anesthesia
Period: Overall Study
Arm/Group | Spinal Anesthesia | General Anesthesia
Started | 91 | 89
Completed | 82 | 80
Not Completed | 9 | 9
Not completed — Protocol Violation | 4 | 8
Not completed — Withdrew consent | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Anesthesia | General Anesthesia | Total
Number analyzed (Participants) | 91 | 89 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 89 | 180
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.9 (5.5) | 46.0 (6.0) | 45.9 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 89 | 180
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 91 | 89 | 180

OUTCOME MEASURES:

1. Primary Outcome: Duration of Hospital Stay.
Description: Duration of hospital stay defined as time from start anesthesia to leaving the hospital
Time Frame: Within 6 months after surgery
Population: Participants who completed the study were analyzed
Measure: Median (Full Range); unit: Hours
Groups:
- Spinal Anesthesia: Spinal anesthesia combined with intrathecal morphine. Spinal anesthesia applied in intervertebral space L3/L4 or L2/L3 with hyperbaric bupivacaine 20 mg and morphine 0.2 mg intrathecally. Sedation with propofol.
- General Anesthesia: General anesthesia. General anesthesia induced with propofol, fentanyl and rocuronium, and maintained with propofol and oxygen in air. Rocuronium and fentanyl repeated when needed.
Arm/Group | Spinal Anesthesia | General Anesthesia
Number analyzed (Participants) | 82 | 80
Hours | 46 [22 to 125] | 50 [24 to 100]

2. Secondary Outcome: Occurrence and Degree of Postoperative Symptoms.
Time Frame: Within 6 months after the surgery
Reporting Status: Not Posted

3. Secondary Outcome: Postoperative Consumption of Analgesics and Antiemetics.
Time Frame: Within 6 months after surgery
Reporting Status: Not Posted

4. Secondary Outcome: Complications and Complication Rates.
Time Frame: Within 6 months after the surgery
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Life and QALYs (Quality Adjusted Life Years).
Time Frame: Within 6 months after the surgery
Reporting Status: Not Posted

6. Secondary Outcome: Sick Leave.
Time Frame: Within 6 months after the surgery
Reporting Status: Not Posted

7. Secondary Outcome: The Stress Coping Ability Impact on Postoperative Symptoms and Recovery.
Time Frame: Within 6 months after the surgery
Reporting Status: Not Posted

8. Secondary Outcome: Health-related Economy.
Time Frame: Within 6 months after the surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Spinal Anesthesia | General Anesthesia
Serious Adverse Events (participants affected / at risk) | 7/91 | 10/89
Other Adverse Events (participants affected / at risk) | 17/91 | 16/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Anesthesia (N=91) | General Anesthesia (N=89)
Urinary bladder injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Infections (Infections and infestations) | 7 (7) | 9 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Anesthesia (N=91) | General Anesthesia (N=89)
Abdominal wound complication (General disorders) | 12 (12) | 10 (10)
Lower urinary tract infection (Renal and urinary disorders) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No